CLINICAL TRIAL: NCT03021590
Title: Comparison Efficacy of 14-day Concomitant Therapy:Clarithromycin vs.Levofloxacin in Eradication of H.Pylori
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No Participants Enrolled
Sponsor: Damascus Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: G5-17
Record Dates: First submitted 2017-01-05; First posted 2017-01-16 (Estimated); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Helicobacter Pylori Gastrointestinal Tract Infection
Keywords: Helicobacter pylori; Helicobacter Infections; Proton Pump Inhibitors; sequential therapy; Clarithromycin; Tinidazole
MeSH Terms: conditions — Helicobacter Infections | interventions — Clarithromycin; Tablets; Esomeprazole; Amoxicillin; Tinidazole; Levofloxacin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clarithromycin :Concomitant Therapy (Experimental): Amoxicillin 1000 mg Tablets, Clarithromycin 500 mg Tablets , Tinidazole 500 mg Tablets and Esomeprazole 20 mg Capsule each every 12 hours for 14 days all by mouth
  Interventions: Drug: Clarithromycin 500Mg Oral Tablet
- Levofloxacin :Concomitant Therapy (Active Comparator): Levofloxacin 500 mg Tablets Amoxicillin 1000 mg Tablets,Tinidazole 500 mg Tablets and Esomeprazole 20 mg each every 12 hours for 14 days all by mouth
  Interventions: Drug: Levofloxacin 500Mg Oral Tablet

INTERVENTIONS:
Drug: Clarithromycin 500Mg Oral Tablet — Amoxicillin 1000 mg Tablets every 12 hours , Esomeprazole 20 mg Capsule days all
  ,Clarithromycin 500 mg Tablets and Tinidazole 500 mg Tablets every 12 hours for 14 days all by mouth
  Other Names: Esomeprazole 40Mg Capsule; Amoxicillin 1000Mg Capsule; Tinidazole 500Mg Tablet
  Arms: Clarithromycin :Concomitant Therapy
Drug: Levofloxacin 500Mg Oral Tablet — Amoxicillin 1000 mg Tablets , Esomeprazole 20 mg Capsule,Levofloxacin 500 mg Tablets and Tinidazole 500 mg Tablets all every 12 hours for 14 days all by mouth
  Other Names: Esomeprazole 40Mg Capsule; Amoxicillin 1000Mg Capsule; Tinidazole 500Mg Tablet
  Arms: Levofloxacin :Concomitant Therapy

SUMMARY:
Comparison Efficacy of 14-day Concomitant therapy between levofloxacin and Clarithromycin on the Eradication of Helicobacter Pylori in Syrian population

ELIGIBILITY:
Inclusion Criteria:

-Patients are aged greater than 18 years old who have H. pylori infection diagnosed by any of following three methods: I-Positive rapid urease test (CLOtest). II-Histologic evidence of H. pylori by modified Giemsa staining. III-Positive 13C-urea breath test. without prior eradication therapy and are willing to receive therapy.

Exclusion Criteria:

* Children and teenagers aged less than 18 years.
* Previous eradication treatment for H. pylori.
* Patients who took any drug, which could influence the study results such as proton pump inhibitor, H2 blocker, mucosal protective agent and antibiotics.
* History of gastrectomy.
* Gastric malignancy, including adenocarcinoma and lymphoma,
* Previous allergic reaction to antibiotics (Amoxicillin, Tinidazole , Levofloxacin) and prompt pump inhibitors (Es-omeprazole).
* Contraindication to treatment drugs.
* Pregnant or lactating women.
* Severe concurrent disease. Liver cirrhosis. Chronic kidney disease.
* Patients who cannot give informed consent by himself or herself.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Helicobacter pylori Eradication rate | 6 weeks after eradication therapy
  Eradication rate according to Intention to treat (ITT) and per-protocol (PP) analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Damascus Hospital, Damascus, Syria

IPD SHARING:
Plan to Share IPD: Undecided